CLINICAL TRIAL: NCT06722807
Title: ClAmpless, Sutureless PartIAl Nephrectomy for Renal Masses (CASPIAN)
Brief Title: ClAmpless, Sutureless PartIAl Nephrectomy for Renal Masses
Acronym: CASPIAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF-GU-011; IRB202500072 (Other: University of Florida)
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Renal Cell Carcinoma (RCC)
Keywords: partial nephrectomy; renal hilar clamping; renal masses; sutureless; clampless; kidney
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clampless, sutureless robotic partial nephrectomy (Experimental)
  Interventions: Procedure: sutureless, clampless partial nephrectomy

INTERVENTIONS:
Procedure: sutureless, clampless partial nephrectomy — All subjects will undergo a clampless, sutureless robotic partial nephrectomy.

SUMMARY:
During partial nephrectomy surgery, efforts at minimizing ischemia while maximizing renal parenchymal volume are desirable to preserve renal function1,2. Not only clamping of the hilum but the renorrhaphy portion of the procedure also can have a significant negative impact on renal function3-5. It is possible to perform this procedure without clamping the hilum and also without formal renorrhaphy. However robust prospective formal evaluation of safety, risks, and potential benefits and whether or not the technique can be employed in a generalized fashion has not been studied.

Demonstration of safety and generalizability may open a whole new avenue of approaching nephron sparing and renal function sparing kidney surgery and decrease potential risks for long term kidney disease in patients with renal masses. This study will investigate the safety, efficacy, and generalizability of the use of clampless, sutureless partial nephrectomy in the treatment of renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age.
* Patients undergoing partial nephrectomy for renal masses ≤ 7 cm
* Subjects must not have more than one active malignancy at the time of enrollment. (Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen [as determined by the treating physician or approved by the Principal Investigator] may be included).
* A clinical diagnosis consistent with renal cell carcinoma, cT1-3 N0 M0 without renal vein thrombus.
* Adequate laboratory test results, including:

  1. Platelets > 50,000/µL
  2. Hemoglobin > 9.0 g/dL
* Written informed consent obtained from the subject and the subject agrees to comply with all the study-related procedures.
* Subjects of childbearing potential (SOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for at least 2 weeks after surgery to minimize the risk of pregnancy. Prior to study enrollment, subjects of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.
* Subjects with partners of child-bearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for 2 weeks following surgery.

Exclusion Criteria:

* Bleeding disorder (any congenital bleeding diathesis)
* Liver dysfunction with end stage liver disease as determined by the treating investigator
* Presence of renal vein thrombus
* End stage renal disease (eGFR < 15 using Cockcroft-gault formula or receiving renal replacement therapy (i.e. dialysis))
* Subjects of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 2 weeks after surgery.
* Subjects who are confirmed to be pregnant or breastfeeding.
* History of any other disease, metabolic dysfunction, clinical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician.
* Prisoners or subjects who are involuntarily incarcerated, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Positive margin rate | 2-3 weeks post-surgery
  Determine the positive margin rate, as measured on the pathology report 2-3 weeks post-surgery.
Transfusion rate | 4 weeks post-surgery
  Determine the transfusion rate, as measured approximately 4 weeks post-surgery via review of patient medical records.

SECONDARY OUTCOMES:
Renal dysfunction (1 day post-surgery) | 1 day post-surgery
  Determine subject renal dysfunction, measured using estimated glomerular filtration rate using Cockcroft-gault formula, at 1-day post-surgery.
Renal dysfunction (2-3 weeks post-surgery) | 2-3 weeks post-surgery
  Determine subject renal dysfunction, measured using estimated glomerular filtration rate using Cockcroft-gault formula, at 2-3 weeks post-surgery.
Renal dysfunction (6 months post-surgery) | 6 months post-surgery
  Determine subject renal dysfunction, measured using estimated glomerular filtration rate using Cockcroft-gault formula, at 6 months post-surgery.
Estimated blood loss | at time of partial nephrectomy
  Determine the estimated blood loss, as determined on the operative report.
Need for ischemia | at time of partial nephrectomy
  Determine how many subjects have a need for ischemia, as determined by need to clamp or not.

CONTACTS AND LOCATIONS:
Overall Officials: Padraic O'Malley, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States